CLINICAL TRIAL: NCT02942849
Title: Prospective Observational Post-Authorisation Study on the Use of Bemfola® in Human Assisted Reproductive Technology
Brief Title: Post-Authorisation Study on the Use of Bemfola® in Human Assisted Reproductive Technology
Status: Completed | Type: Observational
Sponsor: Finox AG (Industry)
Responsible Party: Sponsor
Other Study IDs: FIN-BEM-2016-04
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Infertility
Keywords: Bemfola; r-hFSH; Oocytes; Pregnancy; OHSS
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: r-hFSH — As per standard clinical practice
  Other Names: Bemfola

SUMMARY:
Prospective, non-comparative, multi-centre, multi-country, observational post-authorization study, to correlate predictive factors with number of oocytes in relation to the gonadotropin dose administered using a new r-hFSH product (Bemfola®) for ovarian stimulation and GnRH-antagonists for pituitary suppression

DETAILED DESCRIPTION:
This will be a prospective, non-comparative, multi-centre, multi-country, observational post-authorization study in Germany and Austria. The study will evaluate the use of follitropin alfa (Bemfola®) in controlled ovarian stimulation for IVF/ICSI.

About 30 ART centres will be involved in the study. Upon site initiation, each investigator site will enrol the subjects who meet the inclusion criteria.

As this is an observational study, there will be no additional treatment or diagnostic procedures performed on subjects other than those of the investigators' local routine clinical practice. The decision to start ART treatment and to use Bemfola® in controlled ovarian hyperstimulation (COH) following a GnRH antagonist protocol will be made independently by the investigators as per the ART centre's protocol, preceding patient enrollment for this study.

ELIGIBILITY:
Inclusion Criteria:

* Female subject justifying an IVF/ICSI treatment
* Age over 18 years (inclusive) at the time of the screening visit
* Signed informed patient consent
* Received only Bemfola® for ovarian stimulation
* Pituitary suppression with GnRH-antagonists

Exclusion Criteria:

* Hypersensitivity to the active substance follitropin alfa, FSH or to any of the excipients
* Tumours of the hypothalamus or pituitary gland
* Ovarian enlargement or ovarian cyst not due to polycystic ovarian syndrome
* Gynaecological haemorrhages of unknown aetiology
* Ovarian, uterine or mammary carcinoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise 1800 women intending to undergo ovarian stimulation with Bemfola® in order to have follicular puncture and oocyte retrieval performed as part of an in vitro fertilisation cycle with or without intracytoplasmic sperm injection, for reproductive purposes, and who are pituitary-suppressed with a GnRH antagonist.
  About 30 Fertility centres will be involved in the study. Upon site initiation, each investigator site will enrol the subjects who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1195 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | 34-36 hours after hCG administration

SECONDARY OUTCOMES:
Antral Follicle Count (AFC) | Day 1
Basal FSH level | Day 1
r-hFSH dose on first and last day of stimulation | Day 1 of stimulation through to maximum Day 16 of stimulation
Days of FSH stimulation (with r-hFSH daily doses) | Day 1 of stimulation through to maximum Day 16 of stimulation
r-hFSH total dose | Day 1 of stimulation through to maximum Day 16 of stimulation
Type of oocyte trigger (ß-hCG / GnRH agonist) | At Day of hCG administration
Number of oocytes fertilized (classified as 2PN stages) | Day 1,2,3 or 5 after ovum pick-up/fertilisation
Number of 2PN cells cryopreserved | Day 1,2,3 or 5 after ovum pick-up/fertilisation
Number of embryos transferred | Day 2-5 after ovum pick-up
Proportion of Biochemical pregnancies (determined by serum B-hCG levels) | 15-20 days after oocyte retrieval
Implantation rate (gestational sacs with heartbeat per total number of embryos transferred) | 15-20 days after oocyte retrieval
Incidence of Ovarian Hyper-Stimulation Syndrome (OHSS), classified as mild, moderate and severe | From Day 1 of stimulation
Incidence of ALL other Treatment-Emergent Adverse Events | From Day 1 of study period
Proportion of clinical pregnancies (determined by the presence of a gestational sac) | 35-42 days after oocyte retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Steffen Krüssel, MD, Principal Investigator — Leiter universitäres interdisziplinäres Kinderwunschzentrum Düsseldorf (UniKiD)
Locations (1):
- Team Kinderwunsch Oldenburg, Oldenburg, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided